CLINICAL TRIAL: NCT06301932
Title: The Effectiveness and Outcomes of Epidural Analgesia in Patients Undergoing Open Hepatectomy: A Propensity Score Matching Analysis
Brief Title: The Effectiveness and Outcomes of Epidural Analgesia in Patients Undergoing Open Hepatectomy
Status: Completed | Type: Observational
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Isarapong Pianngarn, Principal Investigator, Chiang Mai University
Other Study IDs: ANE-2562-06771
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Epidural Analgesia; Patient Controlled Analgesia
Keywords: Liver resection; Propensity score matching

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Epidural analgesia: Group of the patients received epidural analgesia
  Interventions: Procedure: Open liver resection
- Non epidural analgesia: Group of the patients who did not received epidural analgesia
  Interventions: Procedure: Open liver resection

INTERVENTIONS:
Procedure: Open liver resection — The definitions of liver resection and the type of hepatectomy were aligned with the anatomic classification of the Brisbane 2000 Terminology

SUMMARY:
This observational study is to compare the effectiveness and outcomes of epidural analgesia in patients undergoing open hepatectomy: A propensity score matching analysis.

The main question is: What is the superior method of pain control in open hepatectomy: epidural analgesia or intravenous PCA?

DETAILED DESCRIPTION:
After approval of the study protocol from the institutional review board of Chiangmai University (Approval number: ANE-2562-06771), the investigators performed a retrospective review of all patients who underwent an elective open liver resection in the specialized hepato-biliary center from January 2007 through December 2018. This retrospective inquiry comprised 612 patients. The data was systematically retrieved from electronic medical records. Baseline characteristics including age, gender, body mass index (BMI), co-morbidity, American Society of Anesthesiologists (ASA) classification, diagnosis, hepatitis profile, Child-Pugh classification, cirrhosis, the largest tumor size, previous liver resection, and pre-operative laboratory investigations were collected. The following intra-operative data were collected: type of liver resection, hilar resection, vascular reconstruction, intra-operative opioid consumption and type of fluid administration, estimated blood loss, packed red cell and blood product transfusion, and operation time. Post-operative pain score and opioid consumption also be collected.

ELIGIBILITY:
Inclusion Criteria:

* All gender age above 18 years old
* Undergoing open liver resection surgery

Exclusion Criteria:

* No documentation of the numerical rating scale (NRS)
* Epidural failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients more than 18 years old, who underwent an open hepatectomy between January 2007 - December 2018 at Maharay Nakhon Chiangmai Hospital
Sampling Method: Non-Probability Sample
Enrollment: 654 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Post-operative opioid consumption | Within 72 hours
  Post-operative opioid consumption at 24,48,72 hour

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pianngarn I, Lapisatepun W, Kulpanun M, Chotirosniramit A, Junrungsee S, Lapisatepun W. The effectiveness and outcomes of epidural analgesia in patients undergoing open liver resection: a propensity score matching analysis. BMC Anesthesiol. 2024 Sep 2;24(1):305. doi: 10.1186/s12871-024-02697-1. PMID 39223470